CLINICAL TRIAL: NCT03015857
Title: A Comparison Between Phenylephrine and Norepinephrine Boluses in Prevention of Post-spinal Hypotension During Cesarean Delivery
Brief Title: Phenylephrine and Noradrenaline for Post Spinal Anesthesia Hypotension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, ahmed elsakka, Principal investigator and lecturer of anesthesia, faculty of medicine cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: cesarean sections
Record Dates: First submitted 2016-12-05; First posted 2017-01-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Adverse Anesthesia Outcome
MeSH Terms: interventions — Phenylephrine; Norepinephrine; Bupivacaine; Fentanyl; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- phenylephrine, (Active Comparator): - Phenylephrine group (n=100): will receive 100 mcg phenylephrine as a single bolus just after intrathecal injection of 10 mg bupivacaine plus 20 mcg fentanyl. The dose will be diluted in 5 mL and given over seconds. A continuous infusion with placebo (normal saline) will start after the first bolus.
  Interventions: Drug: phenylephrine; Drug: Bupivacaine; Drug: Fentanyl; Drug: Placebo (normal saline)
- norepinephrine (Active Comparator): - Norepinephrine group (n=100): will receive bolus of norepinephrine (10 mcg) directly after spinal block using 10 mg bupivacaine plus 20 mcg fentantanyl followed by continuous infusion of norepinephrine with a rate of 0.1 mcg/kg/min till delivery of the fetus.
  Interventions: Drug: Norepinephrine; Drug: Bupivacaine; Drug: Fentanyl

INTERVENTIONS:
Drug: phenylephrine — - phenylephrine; a vasopressor drug given to prevent post spinal hypotension
  Arms: phenylephrine,
Drug: Norepinephrine — - norepinephrine; a vasopressor drug given to prevent post spinal hypotension
  Arms: norepinephrine
Drug: Bupivacaine — intrathecal bupivacaine 10 mg will be given in both groups
Drug: Fentanyl — intrathecal fentanyl 20 mcg will be given in both groups
Drug: Placebo (normal saline)
  Arms: phenylephrine,

SUMMARY:
Hypotension following spinal anesthesia for cesarean section is a serious problem. In this study we investigated the effect of the vasopressors phenylephrine and noradrenaline on postspinal hypotension.

DETAILED DESCRIPTION:
On arrival to the operating room, an 18g cannula will be inserted and monitors will be applied (electrocardiography - pulse oximetry - non-invasive blood pressure monitor). Patients will receive spinal anesthesia with 500 ml rapid crystalloid co-load. Ten milligrams heavy bupivacaine in addition to 20 mcg fentanyl will be injected in L3-L4 or L4-L5 interspace using 25 g spinal needle in the sitting position.

After spinal block, patients will be randomly allocated into one of two groups:

* Phenylephrine group (n=100)
* Norepinephrine group (n=100)

Patients who shows SBP above 140 mmHg or heart rate below 55 bpm after the first vasopressor dose will not receive the infusion. The infusion will stop if the SBP was above 140 mmHg or if the heart rate was below 55 bpm. Patients will be positioned in the supine position with left lateral tilt. Block success will be assessed using pinprick, patients with failed block will be excluded from the study. The highest sensory block level will be assessed after 5 minutes from intrathecal injection. Co-hydration will be continued till maximum of 1.5 litres.

ELIGIBILITY:
Inclusion Criteria:

* full term singleton parturients
* elective cesarean sections

Exclusion Criteria:

* cardiac morbidities
* hypertensive disorders of pregnancy
* peripartum bleeding
* body mass index > 35 will be excluded from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Incidence of post spinal hypotension (PSH) defined as percentage of patients with decreased systolic blood pressure less than 80% of the baseline reading during the period from intrathecal injection to delivery of the fetus) | 2 hours

SECONDARY OUTCOMES:
systolic and diastolic blood pressures measured in mm Hg | 2 hours
heart rate measured in beats per minute | 2 hours
nausea and vomiting measured in number of attacks | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Refaat, M.D., Study Chair — Lecturer of anesthesia Faculty of medicine Cairo university; Tamer M Rook, M.D., Study Chair — Lecturer of anesthesia Faculty of medicine Cairo university

IPD SHARING:
Plan to Share IPD: Undecided